CLINICAL TRIAL: NCT07393152
Title: Studio Pilota su Strumenti Collaborativi, Globali, Multidimensionali e di qualità Della Vita Per la Definizione Delle priorità, lo Sviluppo di Processi Decisionali Condivisi, la Valutazione Degli Esiti e il Miglioramento Della qualità Delle Cure Per le Persone Con Disturbi Dello Spettro Autistico (ASD) Nella Pratica Clinica Quotidiana.
Brief Title: Pilot Study on Collaborative, Comprehensive, Multidimensional and Quality of Life Tools for Priority Definition, Shared Decision Making, Outcome Evaluation and Quality of Care Improvement in ASD Individuals and Programs in the Real World.
Acronym: ASD Outcome
Status: Recruiting | Type: Observational
Sponsor: Antonella Costantino (Other)
Collaborators: IRCCS Eugenio Medea (Other); ASST Valle Olona (Unknown)
Responsible Party: Sponsor-Investigator, Antonella Costantino, Director Child and Adolescence Neuropsychiatric Unit, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico , Milan, Italy, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Organization: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Other Study IDs: 573_12.03.2025_P_bis
Record Dates: First submitted 2025-07-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorders
Keywords: Global functioning; Quality of life; Child and adolescent need and strenght; autism spectrum disorders; Outcome evaluation tools
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged 0-11 with ASD diagnosis: Patients will be enrolled in ongoing treatments in the real context as long as they are in line with the national guidelines for autism, in at least three different national health facilities (SSN) in Lombardy, to represent the variability of the possible organizations of services and interventions, adding new outcome tools.
  Interventions: Other: DD-CGAS (Wagner et al. 2007); Other: Pediatric Quality of Life Inventory (PedsQL).; Other: Child and Adolescent Needs and Strengths (CANS) (Lyons 2022)

INTERVENTIONS:
Other: DD-CGAS (Wagner et al. 2007) — The DD-CGAS is a clinician-completed scale that provides a global rating of the child's functioning. The score refers to the subject's typical functioning during a specified period of time, usually the week prior to the assessment. It is a global assessment based on all available sources of information and all domains of functioning, including self-sufficiency, communication, social behavior, and academic/school functioning. The score should not be influenced by the specific diagnosis, the perceived cause of dysfunction (e.g., cognitive or physical limitation, environmental constraints, behavioral disturbance), or the type and severity of symptoms. The DD-CGAS is a dimensional scale with scores ranging from 1 to 100, with 1 representing the greatest impairment in functioning and 100 representing the best functioning. Each decile (e.g., 1-10, 11-20) has a specific description. The instrument has excellent replicability between raters and temporal stability.
Other: Pediatric Quality of Life Inventory (PedsQL). — The PedsQL is designed for children and adolescents between the ages of 2 and 18 years and takes approximately 5 minutes to complete. It is administered as a self-report instrument or via proxy interview. The proxy interview version corresponds to the age of the child (e.g., 2-4 years, 5-7 years, 8-12 years, and 13-18 years). The PedsQL consists of 23 items that assess 4 broad scales, including: physical functioning, emotional functioning, social functioning, and academic functioning. Items are rated using a 5-point Likert scale (0 = never; 4 = almost always), with the total score calculated as the sum of all items considered. PedsQL item scores are inverted and linearly transformed to a 0 to 100 scale, with higher scores indicating a better perception of health-related quality of life. It is important to note that the PedsQL has been validated in children with autism, including parents of children with autism (Vasilopoulou et al. 2016; Perry, N. et al. 2024).
Other: Child and Adolescent Needs and Strengths (CANS) (Lyons 2022) — The Child and Adolescent Needs and Strengths scale (CANS) (Lyons 2022) is an open source tool widely used to assess the needs and strengths of children, adolescents, and their families, in clinical, educational and social services settings. It is organized into multiple domains that cover various aspects of a child's life. Common domains include life functioning, behavioral/emotional needs, risk behaviors, strengths, caregiver needs and strengths. Additional modules as trauma can be used.The tool uses a scoring system that reflects the level of need or strength in each area. Typically, needs are rated on a scale from 0 to 3, where 0: No evidence of problems; 1: Watchful waiting, preventive action needed; 2: Action or intervention is required; 3: Immediate or intensive action required. Strengths are rated similarly, with higher scores reflecting greater need for action to support the development of each specific strength.

SUMMARY:
ASD is a very complex and lifelong disorder. Patients' functioning is influenced by multiple factors, including treatments, inclusion and life contexts. Nonetheless, outcome measures are still point-specific and highly fragmented, rarely considering global or multidimensional functioning, development or long-term modifications, especially in the real world. The present study considers ongoing real-life treatments in three different NHS settings, in line with the Italian Guidelines. Two age classes will be considered, 0-5 and 6-11, adding new outcome tools pre-post intervention to those already used, to evaluate quality of life, global functioning, multidimensional needs and strengths and shared decision making. Correlations between the different outcome tools will be explored, and possible clusters will be investigated. Acceptability of the outcome tools for the operators, patients and families, as well as usefulness and sustainability in daily practice, will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* ASD diagnosis according to the criteria shared by the regional NFA network
* Age under 12
* Consent from the person holding parental responsibility for health choices

Exclusion Criteria:

* Subjects aged 12 years or older at the time of enrollment
* No consent from the person holding parental responsibility for health choices

Ages: 0 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with ASD enrolled in one of the intervention programs in line with the national guidelines, within the partner institutions or other NPIA/rehabilitation services for developmental age of the Lombardy Region are eligible. The overall expected sample is 400 male and female children, under 12 years of age, 200 children aged 0-5 years at T0 and 200 children aged 6-11 years at T0.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Specific clusters of CANS items that differentiate the profiles of needs and strengths of users at T0. | From March 2025 to August 2026
  The primary objective of the study is to identify specific clusters of CANS items that differentiate the profiles of needs and strengths of users at T0.

SECONDARY OUTCOMES:
Correlations between CANS assessment and participants' global functioning (DD-CGAS) | From March 2025 to August 2026
  The outcome measure TAI measured with CANS and expressed as the sum of the actionable items (see section "Groups and Intervention") will be correlated will be correlated with outcome measure quality of life, measured with DD-CGAS expressed as 1-100 score con 1 che rappresenta la maggiore compromissione del funzionamento e 100 il miglior funzionamento
Correlations between CANS assessment and participants' quality of life (PEDSQL) | From March 2025 to August 2026
  The outcome measure TAI measured with CANS and expressed as the sum of the actionable items (see section "Groups and Intervention") will be correlated will be correlated with outcome measure quality of life, measured with DD-CGAS expressed as 0-100 score with higher scores on the PedsQL indicating better perceptions of health-related quality of life.
Evaluation of changes in children's needs over time based on CANS actionable items. | march 2025 to august 2026
  Differences between T0 and T1 TAI measeured with CANS and expressed as the sum of the actionable items (see section "Groups and Interventions") will be evaluated using a paired sample t test.
Evaluation of changes in children's Quality of Life over time. | from march 2025 to august 2026
  Differences between T0 and T1 PedsQL scores (range 0-100, where 0 represents the lowest quality of life and 100 represents the highest quality of life ) will be evaluated using a paired sample t test.
Evaluation of changes in children's global functioning | from march 2025 to august 2026
  DESCRIPTION Differences between T0 and T1 DD-CGAS scores (range 1-100, where 1 represents the lowest level of global functioning and 100 represents the highest level of global functioning) will be evaluated using a paired sample t test.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - IRCCS Eugenio Medea- U.O. di Neuropsichiatria infantile - Disturbi del Neurosviluppo, Bosisio Parini, (LC)
  - UOSD Disturbo Autistico nel ciclo della vita, Busto Arsizio, (VA)
  - SC Child and Adolescence Neuropsychiatric Unit, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico , Milan, Italy, Milan, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandbank M, Pustejovsky JE, Bottema-Beutel K, Caldwell N, Feldman JI, Crowley LaPoint S, Woynaroski T. Determining Associations Between Intervention Amount and Outcomes for Young Autistic Children: A Meta-Analysis. JAMA Pediatr. 2024 Aug 1;178(8):763-773. doi: 10.1001/jamapediatrics.2024.1832. PMID 38913359
- [Background] Provenzani U, Fusar-Poli L, Brondino N, Damiani S, Vercesi M, Meyer N, Rocchetti M, Politi P. What are we targeting when we treat autism spectrum disorder? A systematic review of 406 clinical trials. Autism. 2020 Feb;24(2):274-284. doi: 10.1177/1362361319854641. Epub 2019 Jul 3. PMID 31269800
- [Background] Perry N, Boulton KA, Hodge A, Ong N, Phillips N, Howard K, Raghunandan R, Silove N, Guastella AJ. A psychometric investigation of health-related quality of life measures for paediatric neurodevelopment assessment: Reliability and concurrent validity of the PEDS-QL, CHU-9D, and the EQ-5D-Y. Autism Res. 2024 May;17(5):972-988. doi: 10.1002/aur.3127. Epub 2024 Apr 10. PMID 38597587
- [Background] Ne'eman A. When Disability Is Defined by Behavior, Outcome Measures Should Not Promote "Passing". AMA J Ethics. 2021 Jul 1;23(7):E569-575. doi: 10.1001/amajethics.2021.569. PMID 34351268
- [Background] Jolliffe, I. T. (2002). Principal Component Analysis (2nd ed.). Springer.
- [Background] Godoy PBG, Sumiya FM, Seda L, Shephard E. A systematic review of observational, naturalistic, and neurophysiological outcome measures of nonpharmacological interventions for autism. Braz J Psychiatry. 2022 Nov 5;44(5):532-547. doi: 10.47626/1516-4446-2021-2222. Epub 2022 Jun 24. PMID 35751600
- [Background] Cordell, K. D. et al. (2016). Patterns and priorities of service need identified through the Child and Adolescent Needs and Strengths (CANS) assessment. Children and Youth Services Review, 60, 129-135.
- [Background] Brown, C. C., Wang, E. W., & Goad, C. (2022). A review of the psychometric properties of the child and adolescent needs and strengths (CANS): Perspectives on the present state of the literature and future directions. Residential Treatment for Children & Youth, 39(3), 331-346.
- [Background] Benzoni, S. et al. (2020). Partecipazione e valutazione di esito nella salute mentale in età evolutiva: gli strumenti della famiglia CANS nell'esperienza italiana. Erickson
- [Background] Babamoradi H, van den Berg F, Rinnan A. Confidence limits for contribution plots in multivariate statistical process control using bootstrap estimates. Anal Chim Acta. 2016 Feb 18;908:75-84. doi: 10.1016/j.aca.2016.01.002. Epub 2016 Jan 7. PMID 26826689